CLINICAL TRIAL: NCT02778841
Title: Comparative Effects of Kinect Game ™ Exercise, Conventional Balance Exercise, and Concurrent Exercise On Knee Proprioception, Balance, And Functional Mobility on Males Elderly
Brief Title: Effects of Exergame, Conventional Exercise, and Mixed Exercise On Proprioception, Balance, & Mobility on Males Elderly
Acronym: FITT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hassan Sadeghi, PhD Student, Institute of Gerontology, University Putra Malaysia, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FPSK(EX14)P031(FR14)
Record Dates: First submitted 2015-12-17; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Accidental Falls
MeSH Terms: interventions — Exercise; Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- XBox Kinact Exercise (Experimental): Kinact game intervention group performed three times per week on non-consecutive days for eight weeks
  Interventions: Other: Exercise
- conventional balance exercises (Experimental): conventional balance exercises group performed three times per week on non-consecutive days for eight weeks
  Interventions: Other: Exercise
- concurrent exercise group (Experimental): Concurrent group performed mixed conventional balance and Xbox Kinact exercises three times per week on non-consecutive days for eight weeks
  Interventions: Other: Exercise
- control Group (No Intervention): There is no exercise for this group

INTERVENTIONS:
Other: Exercise — This study is designed to examine and comparing there intervention program on balance, mobility and knee proprioception among male elderly
  Other Names: Exercise or intervention
  Arms: XBox Kinact Exercise; concurrent exercise group; conventional balance exercises

SUMMARY:
Falling of the elderly as one of the greatest issues and major health problems among the elderly population has produced a further discussion among gerontologists and physical therapists. Moreover, they are considered as one of the major health problems among the aging population and by now around a third of 65-year-old adults fall as a minimum once a year while 6% of such falls cause fractures. Loss of the balance is the main reason for falling among the elderly. Proprioception is the sensory feedback regarding the joint position sense and movement which can accordingly lead to a decrease in the postural stability and steadiness of the elderly people. Proprioception has shown to be a risk factor for falls in older people. proprioception can be modified by physical training. Recently, exergaming, the playing of video games with body movements, has been proposed as effective strategy to deliver exercise.

Aim of study: the current research investigates the effect of 8 weeks videogame game exercise, conventional balance exercise, and a combined of the two (mixed training) on knee proprioception, static balance, and mobility of elderly male. Methodology: The study was designed as a single-blinded, randomized, controlled intervention trial. Sixty-four male ages 65 years and above were randomly assigned into an exergame group, a traditional balance exercise group, a mixed training group or a passive control group. After pretest all participant perform 8 weeks of exercise and measured the effects of the training regimens on proprioception and other functional outcomes as well as mood states in healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be 65 years old and above.
2. The participants should be able to walk independently for a minimum of 10 meter.
3. The participants should be able to do their daily activities such as eating, going to bathroom, and taking a shower.
4. The participants should be able to do low-level balance exercise

Exclusion Criteria:

1. The participants who had cognitive problems.
2. The participants who could not walk and do their daily activities independently.
3. The participants who have knee fracture or joint replacement.
4. The participant who had regular balance exercise or resistance training in lower body in past 3 months.
5. The participant who had neurological and cardiovascular problem

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
knee joint position sense | At Eight weeks
  A Biodex Isokinetic Dynamometer (Biodex 3, 20 Ramsay Rode, Shirley, New York) was used to assess the proprioception of the subjects. The knee joint proprioception was investigated at target angles 30°, 45° and 60° . participants' legs were passively moved to the target angles, their knees were held at the target position for 10 seconds, and then returned to the starting position (90˚). Then, the participants were asked to extend their knees by pushing the dynamometer lever arm toward the previously selected target angle. The mean joint positioning error of the three measurement degrees of error from the target
One Leg stance | At eight weeks
  The single leg stance test or one leg stance (OLS) test was conducted to measure static balance . This test was performed in open and close eye on separate trials.

SECONDARY OUTCOMES:
Time Up and Go Test (TUG) | At Eight Weeks
  Time Up and Go Test, were conducted to measure functional mobility before and after exercise protocol
10 meter walking test | At Eight Weeks
  10 meter walking test was used to measure functional mobility before and after exercise protocol.

IPD SHARING:
Plan to Share IPD: No
I am not prefer to share data now

REFERENCES:
- [Derived] Sadeghi H, Jehu DA, Daneshjoo A, Shakoor E, Razeghi M, Amani A, Hakim MN, Yusof A. Effects of 8 Weeks of Balance Training, Virtual Reality Training, and Combined Exercise on Lower Limb Muscle Strength, Balance, and Functional Mobility Among Older Men: A Randomized Controlled Trial. Sports Health. 2021 Nov-Dec;13(6):606-612. doi: 10.1177/1941738120986803. Epub 2021 Feb 13. PMID 33583253